CLINICAL TRIAL: NCT05411848
Title: Evaluation of a Nutritionally Complete, Plant-based, High Energy, High Protein, Enteral Tube Feed in Adults
Brief Title: 2kcal Tube Feed Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2KCAL2022
Record Dates: First submitted 2022-05-18; First posted 2022-06-09 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Enteral Nutrition; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Patients will receive a minimum of 1 bottle per day of either (or both of) 2kcal HP PlantBased and/or 2kcal HP PlantBased MultiFibre Tube Feeds for a minimum of 7 days and a maximum of 28 days. During the 12-month follow-up, patients will have access to the same trial prescription as per the 28-day intervention period.
  Interventions: Dietary Supplement: 2kcal HP PlantBased

INTERVENTIONS:
Dietary Supplement: 2kcal HP PlantBased — Patients will receive a minimum of 1 bottle per day of either (or both of) 2kcal HP PlantBased and/or 2kcal HP PlantBased MultiFibre Tube Feeds for a minimum of 7 days and a maximum of 28 days. During the 12-month follow-up, patients will have access to the same trial prescription as per the 28-day intervention period.

SUMMARY:
The primary aim of this study is to investigate the effects of a plant-based, high energy, high protein tube feed with and without inclusion of fibre on gastrointestinal tolerance in adult patients who require nutritional support via enteral tube feeding over a 28-day period, followed by a 12-month follow-up. Secondary aims are to determine the effects on compliance, acceptability, anthropometry, nutrient intake, and physical function. This is a prospective, longitudinal, 28-day intervention study with a 1-day baseline period and a 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* ≥16 years of age
* Using or requiring an enteral tube feed in the community as part of nutritional management plan
* Expected to receive at least 1000kcal/day (one bottle) from one of the study products

Exclusion Criteria:

* Receiving parenteral nutrition
* Patients with major hepatic dysfunction (i.e., decompensated liver disease)
* Patients with major renal dysfunction (i.e., requiring filtration or stage 4/5 chronic kidney disease (CKD))
* Patients receiving inpatient care
* Known pregnancy or lactation
* Participation in other clinical intervention studies within 1 month of this study
* Allergy to any study product ingredients
* Investigator concern regarding ability or willingness of patient to comply with the study requirements.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change in gastrointestinal tolerance | Change from baseline (Day 1) to end of intervention (7-28 days)
  A standardised gastrointestinal (GI) tolerance questionnaire to capture perceived severity (none, mild, moderate or severe) of common gastrointestinal symptoms (diarrhoea, constipation, bloating, abdominal discomfort, vomiting and nausea).
Change in gastrointestinal tolerance | Change from baseline (Day 1) to end of follow-up (12 months)
  A standardised gastrointestinal (GI) tolerance questionnaire to capture perceived severity

SECONDARY OUTCOMES:
Acceptability | Baseline to end of intervention (7-28 days) and end of follow-up (12 months)
  Acceptability (e.g., liking, ease of use, preference) will be assessed by a questionnaire. Questions will be rated on a 7-point Likert scale.
Compliance | Baseline to end of intervention (7-28 days) and end of follow-up (12 months)
  Compliance with the study product prescription (%) will be assessed daily by recording how much of the study product was prescribed compared to the amount administered.
Dietary intake | Baseline to end of intervention (7-28 days) and end of follow-up (12 months)
  A 24-h dietary recall will be conducted to record all food, drink and nutritional feeds taken in the 24 hours prior for analysis of of nutritional intake (i.e., total energy and macro- and micronutrients).
Anthropometry | Baseline to end of intervention (7-28 days) and end of follow-up (12 months)
  Body weight (kg) will be measured using standard methods to the nearest 0.1kg using a weighing scale without heavy clothing. Height will be measured at baseline only using standard measures to the nearest 0.1cm, without shoes or socks. . Height and weight measures will be used to calculate body mass index (BMI).
Dietetic goal | Baseline to end of intervention (7-28 days) and end of follow-up (12 months)
  A dietetic goal (e.g., weight increase/maintenance, improved/maintained GI tolerance, improved/maintained compliance) will be set by the investigating dietitian at baseline (Day 1) for each patient. At the end of the intervention period, the investigating dietitian will assess and note if the dietetic goal was met.
Safety (Adverse events) | Baseline to end of intervention (7-28 days) and end of follow-up (12 months)
  Adverse events will be recorded throughout the study
Calf circumference | 6-months to 12-months follow-up
  Calf circumference (of the dominant leg) will be measured using standard measures to the nearest 0.1cm using a measuring tape
Handgrip strength | 6-months to 12-months follow-up
  Dominant handgrip strength (kg) will be assessed using a handgrip dynamometer
30-s Chair Stand Test | 6-months to 12-months follow-up
  Number of times patients can stand up and sit down from a chair as many times as possible within 30 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Nutricia Ltd., Trowbridge, Wiltshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No